CLINICAL TRIAL: NCT06327464
Title: The Effect of Exogenous Ketones on Appetite in Adults With or Without Obesity
Brief Title: Exogenous Ketones and Appetite
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Sarah Purcell, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 23-03228
Record Dates: First submitted 2024-02-23; First posted 2024-03-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Appetite; Obesity; Ketones; Appetitive Behavior
Keywords: appetite; energy expenditure; exogenous ketones; dietary intake
MeSH Terms: conditions — Obesity; Ketosis; Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone supplement condition first (Other)
  Interventions: Dietary Supplement: Exogenous ketones
- Ketone supplement condition second (Other)
  Interventions: Dietary Supplement: Exogenous ketones

INTERVENTIONS:
Dietary Supplement: Exogenous ketones — Consumption of a single exogenous ketone supplement with breakfast

SUMMARY:
People with obesity have different appetitive responses to stimuli compared to people without obesity. For example, people with obesity have a blunted postprandial ghrelin ('hunger' hormone) response, lower glucagon-like peptide 1 (GLP-1) and peptide-YY (PYY; associated with satiety) compared to people without obesity. Given the favorable effects of exogenous ketones on appetite previously observed in healthy adults of normal body weight, it is possible that these supplements can alter appetite hormones in a manner that may closer match that observed in people without obesity. To explore this research question, investigators will conduct a randomized single-blind cross over study to characterize appetite and dietary intake after ingestion of an exogenous ketone supplement within adults with obesity (compared a control condition without exogenous ketones) and compared to adults without obesity. The research team will also explore differences in postprandial energy expenditure and fuel utilization. Twenty-two healthy young- and middle-aged adults will be included (up to n=26 enrolled). In addition to a baseline visit to measure body composition, participants will undergo two 4.5-hour study visits, one of which will include a ketone diol supplement and one will have a placebo. Participants will be given a 1-day run-in diet prior to each study day to support energy balance. On each study day visit, participants will undergo a resting metabolic rate test (indirect calorimetry) followed by a fasting appetite rating and blood sample collection. Participants will then be provided with a standard breakfast meal (one with the ketone supplement and one with placebo). Appetite ratings and blood sample collection will be repeated 60, 120, and 180 minutes after the meal. Indirect calorimetry will be completed after the 30, 90, and 150 minute assessments. After the 180-minute timepoint, participants will be provided with a buffet-like lunch meal with instructions to eat as much or as little as they would like to determine ad libitum dietary intake at a single meal. To assess free-living ad libitum dietary intake, participants will receive 1.5 days of food boxes tailored to their preferences, with uneaten food returned at the end of the 1.5-day period. This study will be the first to assess the impact of exogenous ketones on appetite in obesity and would help inform future weight loss intervention trials.

DETAILED DESCRIPTION:
Overview:

Investigators will conduct a randomized, single-blind cross-over study in adults with and without obesity. The study consists of one screening/baseline visit, plus two 4.5-hour in-lab appetite visits: one with the exogenous ketone supplement and one without. After the baseline/screening visit, individuals will be randomized to either placebo/ketone or ketone/placebo study visit order in a 1:1 manner using online software (http://www.randomization.com). A washout period of at least 7 days will occur between study visits. For females, every attempt will be made to book these visits in the same menstrual cycle phase (according to self-reported menstrual cycle history) or estimated phase (for individuals not taking hormonal contraceptives or with a hormonal IUD).

Screening and baseline visit (~1 hour):

Individuals who consent to enroll in the study will be scheduled for a ~1 hour visit to confirm eligibility, measure body composition, and review study day procedures. Height and weight will be collected to confirm eligibility. Participants will also complete questionnaires to collect data on basic demographics and medical history, menstrual cycle history (for females), food preferences for the run-in and study day diets, screening for disordered eating (EATS-26) and alcohol or drug abuse (CAGE).

Data on participant's fat mass (FM), fat-free mass (FFM), body fat percent and bone mineral density will be collected using a full body dual X-ray absorptiometry (DEXA; Hologic Model A). Body composition variables will be expressed in absolute terms and controlling for height (e.g. FM index: FM [kg]/height [m2]); FFM will also be expressed in relation to FM (FM:FFM).

Run-in energy balanced diet A 1-day energy-balanced run-in diet will be provided to each participant prior to each study day. Diets will be modified according to participant preferences and the same diet will be given on the second run-in day. The caloric value of the diet will be determined using the 2023 dietary reference intake equations with self-identified activity factor (collected at the screening and baseline visit), and will have a macronutrient composition of 50% carbohydrate, 30% fat, and 20% protein. This baseline dietary control period will ensure energy balance and weight maintenance prior to each study day. All meals will be prepared by a third-party dietary meal prep company in Kelowna.

Study visit days (~4.5-5 hours)

Participants will be asked to refrain from food and calorie- or caffeine-containing beverages for at least 12 hours, alcohol for at least 24 hours, and vigorous-intensity exercise for at least 48 hours before each study visit. Each study day visit will be scheduled to start sometime between 7 - 9:30am, depending on scheduling availability and usual participant wake time; both visits will be scheduled at approximately the same time. All study day procedures will be conducted on the first floor of RHS in the following order:

* Body weight on a digital scale, measured without shoes or heavy clothing items
* Resting metabolic rate will be measured for 15-20 minutes after a period of 25-30 minutes of quiet rest using an indirect calorimeter metabolic cart with face mask (ParvoMedics TrueOne 240). This test measures oxygen consumed and to estimate resting metabolic rate (in kilocalories/day). During the test, participants breathe normally through a facemask, while relaxed but not falling asleep.
* The following procedures will be completed after the resting metabolic rate test, but before breakfast (timepoint '-5'; fasted sample) and 60, 120, and 180 minutes after breakfast is consumed:

  * Serial blood sampling: First, a 22-gauge intravenous (IV) catheter will be placed in the antecubital area of the arm or dorsal side of the hand. For each timepoint, two 3-mL tubes (pretreated ethylenediaminetetraacetic acid [EDTA]) labeled with the participant's study ID, study number, date, and time will be collected. 0.6 mg AEBSF inhibitor will be immediately added to one sample and 0 μL Dipeptidyl peptidase-IV inhibitor and 0.05 mL of aprotinin will be added to the other sample. These samples will be immediately placed on ice stored in a -80 freezer until analyses. The following appetite hormones will be assessed: acylated ghrelin, PYY (radioimmunoassay), GLP-1 (7-36), leptin, and insulin (enzyme-linked immunoassay [ELISA]).
  * Circulating concentrations of glucose and D-β-hydroxybutyrate (ketone) concentrations will be collected using a glucose and ketone monitoring system (Fora 6 Connect).
  * Appetite ratings will be completed using visual analogue scale (VAS) questions about hunger, fullness, prospective food consumption, and desire to eat on a sliding scale on a university-owned iPad. Questions will be from Flint et al. (In J Obes 2000; 24:38-48) and are standard procedure in the greater appetite literature.
  * Additional 30-minute assessments of postprandial energy expenditure and fuel utilization will be collected using indirect calorimetry after the 30, 90, and 120-minute time points. Postprandial energy expenditure assessments will be expressed relative to the resting metabolic rate values.
* Standard breakfast meal: Participants will be given a standard breakfast meal consisting of a protein bar, juice, and mixed nuts (or similar substitutes, in case of food intolerances/allergies). The energy content of the breakfast in both conditions (ketone and placebo) will be designed to meet 25% of each individual's estimated total energy requirements (calculated from the 2023 Dietary Reference Intake equations). In the placebo condition, the macronutrient composition of 50% carbohydrate, 30% fat and 20% protein. In the ketone condition, 70 kcal of carbohydrate will be removed from the breakfast and replaced with the 70-kcal Ketone-IQ supplement. Participants will have up to 20 minutes to consume this meal in a private and quiet location and may not use personal devices, computers, or read during this time to avoid the influence of external stimuli on dietary intake.
* Exogenous ketone and placebo supplements will be delivered in liquid form and consumed orally with the breakfast meal. Both drinks will be diluted to 500mL with a commercially available calorie-free drink (Mio; Kraft-Heinz, Chicago, IL). The ketone supplement (R-1,3-butanediol [HVMN Ketone 2.0]) and taste-matched calorie-free placebo will be provided by HVMN.
* Ad libitum dietary intake at a single lunch meal: At the end of the 180-minute time point, participants will be offered a buffet-style lunch with pre-weighed food items, including: pre-packaged spaghetti with sauce (e.g., Stouffers or similar), dinner rolls, butter, fresh fruit, salad or steamed vegetables, cookies, chips, juice, granola bars, and regular and diet soda. Participants will be asked to consume as much or as little as they like, until comfortably full, and can request more of any item. The meal will be consumed in isolation with no distractions or and the use of computers or mobile phones. At the end of the buffet meal, leftover food will be weighed, and absolute energy and macronutrient intake will be determined by calculating the weighed difference of each food item before and after each meal.

Post-study day visit dietary intake assessment

• Ad libitum dietary intake: Participants will be provided with 1.5 days of meals and snacks to begin consuming after the study day visit. Participants will be instructed to eat as little or as much as they would like in free-living settings. Meals will be provided by a local meal delivery service and supplemented with snacks and beverages purchased by the study team. The content of the provided food will be identical between visits and be determined according to participant's reported eating habits, excluding both top-rated foods and disliked ones to avoid over- and under- consumption. Participants will be asked to only eat the food provided and return empty containers and remaining food at the end of the 1.5-day period. They will be provided with a paper form and food scale to record any foods that were consumed that were not provided.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-45 years
* Body mass index (BMI): 18.5 - 40.0 kg/m2
* For females: Premenopausal, with regular menstrual cycle (every 21-38 days, by self-report) OR lack of regular menstrual cycles due to oral contraceptive or intrauterine device (IUD) use
* Sedentary or recreationally active, defined as: <300 minutes per week of voluntary exercise at moderate intensity or greater over the past 12 weeks
* Not currently pregnant or lactating, not planning to become pregnant in the next 12 weeks
* Ability and willingness to fast for 12 hours before each study day visit
* If applicable:

  * For people who occasionally (i.e., <1x/day) use cannabis (including cannabidiol-based products): ability and willingness to abstain from cannabis for two days prior to each study day visit, the day of each study visit, and during each ad libitum diet phase.
  * For people who use cannabis daily: ability and willingness to continue to use the exact same amount of cannabis as they normally use for two days prior to each study day visit, the day of each study visit, and during each ad libitum diet phase.

Exclusion Criteria:

* Current or previous major comorbidities, by self-report, including:

  * Cardiovascular diseases
  * Diabetes (type 1 or type 2)
  * Cancer
  * Thyroid diseases
  * Human immunodeficiency virus or hepatitis B or C
  * Renal diseases
  * Hepatic diseases
  * Polycystic ovary syndrome
* Uncontrolled/untreated (self-report):

  * Hypertension
  * Dyslipidemia
  * Uncontrolled Ssleep disorders (e.g., insomnia)
  * Any other condition that may affect appetite and energy balance
* Currently or in the past six months:

  * Use of regular medication or supplement that may affect appetite, energy balance, or sleep
  * Regular use of tobacco or nicotine products
* Starting any new prescription medication within two weeks of the first study day visit or during the study
* Working night shifts or traveling across more than 2 time zones within two weeks of and throughout the study
* Food intolerances or allergies that cannot be accommodated
* History of surgical procedure for weight loss at any time (e.g., gastroplasty, gastric bypass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve); history of extensive bowel resection for other reasons
* Current alcohol or substance abuse (score >2 on the cut down-annoyed-guilty-eye opener [CAGE] questionnaire16)
* Current or past history of eating disorders including anorexia nervosa, bulimia, binge eating disorder (self-report or score >20 on the Eating Attitudes Test - 26 [EATS-26] questionnaire17)
* Weight loss >5% in past 12 weeks for any reason

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Acylated ghrelin area under the curve (AUC) | 3 hours
  Acylated ghrelin pre-breakfast and 60, 120, and 180 minutes after breakfast

SECONDARY OUTCOMES:
Peptide-YY(3-36) area under the curve (AUC) | 3 hours
  Peptide-YY(3-36) pre-breakfast and 60, 120, and 180 minutes after breakfast
Glucagon-like peptide 1 area under the curve (AUC) | 3 hours
  Glucagon-like peptide 1 pre-breakfast and 60, 120, and 180 minutes after breakfast
Insulin area under the curve (AUC) | 3 hours
  Insulin pre-breakfast and 60, 120, and 180 minutes after breakfast
Glucose area under the curve (AUC) | 3 hours
  Glucose pre-breakfast and 60, 120, and 180 minutes after breakfast
Leptin area under the curve (AUC) | 3 hours
  Leptin pre-breakfast and 60, 120, and 180 minutes after breakfast
Hunger rating from visual analog scale | 3 hours
  Hunger pre-breakfast and 60, 120, and 180 minutes after breakfast (see detailed description)
Satiety rating from visual analog scale | 3 hours
  Satiety pre-breakfast and 60, 120, and 180 minutes after breakfast (see detailed description)
Prospective food consumption rating from visual analog scale | 3 hours
  Prospective food consumption pre-breakfast and 60, 120, and 180 minutes after breakfast (see detailed description)
Desire to eat rating from visual analog scale | 3 hours
  Desire to eat pre-breakfast and 60, 120, and 180 minutes after breakfast (see detailed description)
Dietary energy intake at a single meal | 1 hour
  Ad libitum intake at lunch; difference between energy in weighed food before and after consumption in a laboratory setting
Free-living dietary energy intake | 1.5 days
  Ad libitum intake; difference between energy in weighed food before and after consumption, provided to participants in free-living environments
Postprandial energy expenditure | 3 hours
  Energy expenditure before breakfast and 30, 90, and 150 minutes after breakfast

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia - Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No